CLINICAL TRIAL: NCT02156505
Title: Phase IV Study of Double Bare Self-expandable Metallic Stent for Malignant Gastric Outlet Obstruction
Brief Title: Outcome Study of Double Bare Stent for Malignant Gastric Outlet Obstruction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Stent research group, Korean Society of Gastrointestinal Endoscopy, Korea (Unknown)
Responsible Party: Principal Investigator, Chan Gyoo Kim, Senior scientist, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTSMD12009
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Gastric Outlet Obstruction Due to Malignancy
Keywords: stent; gastric outlet obstruction; restenosis
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DoubleBare stent (Experimental): Placement of double bare stent
  Interventions: Procedure: placement of double bare stent; Device: DoubleBare stent

INTERVENTIONS:
Procedure: placement of double bare stent
Device: DoubleBare stent

SUMMARY:
Self-expandable metallic stents provide effective palliation of malignant gastric outlet obstruction. However, uncovered stent are often associated with re-stenosis caused by tumor in-growth through the stent mesh. The Self-expandable metallic stents which has the design of smaller wire mesh size (double bare stent) were developed and used in Korea. This new design was developed to minimize the re-stenosis of uncovered stent, but the outcome is unknown. The end point of this study is the 8-weeks patency rate after placement of double bare as well as technical and clinical success rates.

ELIGIBILITY:
Inclusion Criteria:

* Malignant gastric outlet obstruction
* Symptoms compatible with gastric outlet obstruction
* An inoperable condition because of extent of disease or patient's conditions

Exclusion Criteria:

* History of enteral stent placement, undergone gastric surgery.
* Additional small bowel stenosis distal to gastric outlet obstruction.
* Refuse to be enrolled to study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The patency rate at 8 weeks after placement. | 8 weeks

SECONDARY OUTCOMES:
Technical and clinical success rates | up to 8 weeks
re-stenosis rate | 8 weeks
migration rate | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea